CLINICAL TRIAL: NCT03486574
Title: Research for Associated Genes for Developing Gastric Cancer in Family Member With First-Degree Relatives of Gastric Cancer
Brief Title: Research for Associated Genes for Gastric Cancer in Family Member With Affected First-Degree Relatives
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1610/366-303
Record Dates: First submitted 2018-03-24; First posted 2018-04-03 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Gastric Cancer; Genetic Predisposition
MeSH Terms: conditions — Stomach Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from 10ml of plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric cancer: Pathologically proven diseases after upper gastroendoscopy and biopsy. Previous pathological reports and endoscopic image can be used.
  Interventions: Diagnostic Test: Positive result from pathological test
- non-gastric cnacer: Rull out gastric cancer by upper gastroendoscopy. The results 3 moths before enrollment is available.

INTERVENTIONS:
Diagnostic Test: Positive result from pathological test — Presence/absence of gastric cancer will be evaluated by upper gastroendoscopy or results of pathological test
  Groups: Gastric cancer

SUMMARY:
Familial gastric cancer accounts for 10% of all cases, but predisposing genetic variations is unknown except for CDH1 mutation.

Because Germline mutation is believed to be a key aspect of cancer predisposition, we plan to recruit persons with 2 or more affected family members in three-generation pedigree. The investigators will perform a whole-exome sequencing using DNA from blood samples of families including gastric cancer patients and non-gastric cancer patients

DETAILED DESCRIPTION:
1> Patient selection

Enroll criteria:

1) Gastric cancer patients and their first-degree relatives and 2) family with two or more gastric cancer patients within three-generation pedigree.

A three-generation pedigree will be used for diagnostic consideration or risk assessment of rare variation.

Personal history will be acquired by questionnaire which asks smoking, alcohol intake, dietary preference, socioeconomic information and history of previous eradication of HP. For any family member with gastric cancer, age at diagnosis, histology type, methods of treatment or pathological reports will be evaluated.

2> Whole exome sequencing, variant annotation, filtering and prioritization After whole exome sequencing, functional annotation of genetic variants will be conducted using ANNOVAR.

3> Linkage analyses To perform variant and gene-based linkage analysis in pedigrees, data will be analyzed using pedigree-VAAST.

4> Validation using a genechip

ELIGIBILITY:
Inclusion Criteria :

* Gastric cancer patients and their first-degree relatives
* Members in family with two or more gastric cancer patients within three- generation pedigree

Exclusion Criteria :

* Those who reject the enrollment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigator will recruit or invite the participants among persons who visit the clinic with a family history of gastric cancer.
  The investigator plans to recruit gastric cancer patients and non-patients in family with 2 or more affected members.
  Non-gastric cancer patients was restricted to persons over 50 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Genes with logarithm of odds (LOD)>2 in linkage analysis | 0 day (baseline)
  Based on LOD at baseline, candidate genes will be selected.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided